CLINICAL TRIAL: NCT05912062
Title: Early On-treatment Transcriptional Profiling as Predictor of Response in Early-stage HER2-positive Breast Cancer (BiOnHER)
Brief Title: Early On-treatment Transcriptional Profiling as Predictor of Response in Early-stage HER2-positive Breast Cancer
Acronym: BiOnHER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundación Sociedad Española de Oncologia Médica (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Reveal Genomics (Registered trademark) (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI20/00544
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: HER2-positive Breast Cancer; Neoplasms; Breast Cancer
Keywords: Neoadjuvant HER2-positive Breast Cancer; Human Epidermal Growth Factor Receptor 2; Biomarker; Radiomic; Transcriptomics; Spatial transcriptomics; HER2Dx
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Trastuzumab; Neoadjuvant Therapy; pertuzumab; Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- early-stage HER2-positive breast cancer neoadjuvant treatment: For a total of 16 weeks, patients will be given dual antiHER2 blockade consisting of Cycle 1 Day 1 Pertuzumab 840mg + Trastuzumab 8mg/kg loading dose, followed by Paclitaxel starting at Cycle 1 day 8 and 15 at 80mg/m2. Followed by Pertuzumab 420mg + Trastuzumab 6mg/kg every three weeks and Paclitaxel days 1, 8, and 15 of a 21-day cycle for up to fifteen weeks.
  Adjuvant treatment (including the need of Anthracyclines) will be administered according clinical practice.
  Interventions: Drug: Trastuzumab (neoadjuvant); Drug: Pertuzumab (neoadjuvant); Drug: Paclitaxel (neoadjuvant)

INTERVENTIONS:
Drug: Trastuzumab (neoadjuvant) — Trastuzumab loading dose at 8mg/kg at day 1 followed by Trastuzumab at 6mg/kg in a 21-day cycle for six cycles
Drug: Pertuzumab (neoadjuvant) — Pertuzumab loading dose at 840mg at day 1 followed by Pertuzumab at 420mg in a 21-day cycle for six cycles
Drug: Paclitaxel (neoadjuvant) — Paclitaxel starting at day 8 at 80mg/m2, days 1, 8, and 15 of a 21-day cycle for up to fifteen weeks

SUMMARY:
Non-randomized, open label, translational research study in women with early HER2-positive invasive breast carcinoma eligible for neoadjuvant treatment.

The aim of BIONHER is to assess the impact of short-term neoadjuvant dual HER2-blockade on HER2-positive breast cancer transcriptomic profile and to evaluate whether early on treatment tumor biopsy can improve the accuracy of predicting response over the pre-treatment alone.

DETAILED DESCRIPTION:
This is a prospective study of paired tumor samples from patients with newly diagnosed HER2-positive breast cancer eligible for neoadjuvant treatment to evaluate whether early on-treatment biomarkers can improve the accuracy of predicting response over pre-treatment samples alone.

Sequential tumor biopsies will be obtained at two time points: before initiation of neoadjuvant dual HER2-blockade (pre-treatment, day 1) and 1 week later (day 8), before introduction of paclitaxel to the neoadjuvant treatment.

Following the completion of neoadjuvant paclitaxel, trastuzumab and pertuzumab (THP) for 16 weeks, patients will proceed to surgery. After surgery, adjuvant treatment (including need for Anthracyclines) will be followed as per clinical practice.

The study will comprise two phases: a discovery phase (n=60) where sequential paired tumor biopsies will be used for RNA-Seq analysis and assessment of tumor infiltrating lymphocytes (TILs) and CelTIL score. Radiomic characteristics of MRI, HER2Dx® and spatial transcriptomics (using GeoMx®) will be also evaluated.

This phase will be followed by a validation phase (n=20) in which prediction accuracy observed in the discovery phase will be validated by Nanostring gene expression analysis using a new cohort of patients with HER2-positive breast cancer eligible for neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning specific protocol procedures
* Untreated invasive breast carcinoma eligible for neoadjuvant treatment
* Histologically or cytologically confirmed human epidermal growth factor receptor 2 positive (HER2) Breast Cancer defined by ASCO/CAP guidelines based on the most recent analyzed biopsy or other pathology specimen; independently for estrogen receptor (ER) and progesterone receptor (PR)
* Female and male patients
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function defined as: Absolute neutrophil count (ANC) ≥1.5 × 109/L, Hemoglobin (Hgb) ≥10 g/dL, Platelets >100 000/mm3, Creatinine ≤1.6 mg/dL, ALT and AST ≤2.5 × ULN, Alkaline phosphatase ≤5 ULN, Total bilirubin ≤1.5 mg/dL
* Baseline LVEF ≥50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan
* Negative β-HCG pregnancy test (serum) for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after the menopause. All subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control from 2 weeks before administration of the first dose of investigational product until 28 days after last dose of investigational product
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Exclusion Criteria:

* Known metastatic disease
* Known or suspected hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances
* Concurrent congestive heart failure or LVEF <50%
* History of significant comorbidities that, in the judgment of the investigator, may interfere with the conduction of the study, the evaluation of response, or with informed consent
* Use of any investigational agent or participation in another therapeutic clinical trial concurrently or in the previous 30 days before the enrollment
* Patients who are pregnant or breast-feeding
* Women of child-bearing potential who are unable or unwilling to use contraceptive measures
* Inability or unwillingness to abide by the study protocol or cooperate fully with the investigator
* Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy other than the trial therapies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in this study will be patients with early-stage HER2-positive breast cancer treated with neoadjuvant trastuzumab, pertuzumab (HP) and paclitaxel within standard clinical practice at the Catalan Institute of Oncology (ICO) Hospitalet.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in gene expression (by RNA-seq technology) induced by a single dose of dual HER2-blockade with pertuzumab and trastuzumab. | Between day 1 and day 8

SECONDARY OUTCOMES:
Gene expression patterns (by RNA-seq technology) induced by a single dose of dual HER2-blockade with pertuzumab and trastuzumab to better predict pathological complete response (pCR) in HER2-positive breast cancer | Between day 1 and day 8
Characterize the immune component of the tumor microenvironment (TME) using Spatial transcriptomics. | Between day 1 and day 8
Changes in the immune component of TME induced early by treatment after the first dose of dual anti-HER2 blockade that are associated with pCR. | Between day 1 and day 8
Clinical and radiomic characteristics of MRI together with machine learning for a better prediction of which patients will achieve a pCR and which will not | Between MRI at diagnosis and pre-surgery
Machine learning for a construction and validation of (by Nanostring technology) an early predictor of response to the neoadjuvant treatment to distinguish between responders and nonresponders. | Between day 1 and day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català d'Oncologia l'Hospitalet, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pernas S, Guerriero JL, Naumenko S, Goel S, Regan MM, Hu J, Harrison BT, Lynce F, Lin NU, Partridge A, Morikawa A, Hutchinson J, Mittendorf EA, Sokolov A, Overmoyer B. Early on-treatment transcriptional profiling as a tool for improving pathological response prediction in HER2-positive inflammatory breast cancer. Ther Adv Med Oncol. 2022 Jul 30;14:17588359221113269. doi: 10.1177/17588359221113269. eCollection 2022. PMID 35923923